CLINICAL TRIAL: NCT06664424
Title: Non-Inferiority Analysis of Adhesive Strips Vs. Sutures in Lumbar Spinal Fusion: a Propensity Matched Retrospective Study
Brief Title: Adhesive Strips Vs Sutures in Skin Closure for Lumbar Spinal Fusion
Status: Completed | Type: Observational
Sponsor: Diakonie-Klinikum Stuttgart (Other)
Responsible Party: Sponsor
Other Study IDs: Diak 002/2024
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Surgical Site Infections; Lumbar Spinal Fusion
Keywords: Lumbar spinal fusion surgery; surgical site infections; sutures; adhesive strips; non-inferiority study; wound infections; superficial wound infections
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adhesive strips group: Patients in whom adhesive strips were employed for skin closure
- Suture group: Patients in whom sutures were employed for skin closure

SUMMARY:
Comparison between two methods for skin closure in lumbar spinal fusion surgery, a non-inferiority approach between sutures and adhesive strips and its effect on surgical site infections.

DETAILED DESCRIPTION:
Surgical site infections (SSIs) are among the most common complications in spine surgery, the average rate of infection in spine surgery has been estimated to be around 2.1-3.1%, being the lumbar region the most prone to infection with a reported incidence of 3.7-6.9%. Wound management and the choice of materials used for skin closure can influence the rate of wound-related complications.

This work is a retrospective, mono-centric analysis of data collected for surgical site infections (SSIs) surveillance in patients with lumbar spinal fusion surgery, the primary outcome is surgical site infections rate in the cohort and its relation to the wound closure method (Adhesive strips vs sutures). Using a propensity score matching and a non-inferiority analysis the objective was to determined if adhesive strips is not inferior to sutures regarding SSIs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal fusion surgery.
* Open posterior approach.
* Surgery involving one or two spinal segments.
* Patients aged 18 years or older.
* Skin closure performed using either sutures or adhesive strips.

Exclusion Criteria:

* History of previous surgical site infections.
* Diagnosis of spondylodiscitis.
* Postoperative complications unrelated to surgical site infections.
* Deep surgical site infections (A3 classification).
* Patients undergoing surgeries other than lumbar spinal fusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of both genders, aged 18 years or older, who underwent lumbar spinal fusion surgery involving one or two segments, with skin closure performed using either sutures or adhesive strips.
Sampling Method: Non-Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Surgical site infections | 30 days
  Surgical site infections suspected by clinical signs, and confirmed by culture.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Santos-Marcial, P.D. Dr. med, Principal Investigator — Diakonie Klinik Stuttgart
Locations (1):
- Diakonie Klinikum Stuttgart, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boody BS, Jenkins TJ, Hashmi SZ, Hsu WK, Patel AA, Savage JW. Surgical Site Infections in Spinal Surgery. J Spinal Disord Tech. 2015 Dec;28(10):352-62. doi: 10.1097/BSD.0000000000000339. PMID 26566255
- [Background] Zempsky WT, Zehrer CL, Lyle CT, Hedbloom EC. Economic comparison of methods of wound closure: wound closure strips vs. sutures and wound adhesives. Int Wound J. 2005 Sep;2(3):272-81. doi: 10.1111/j.1742-4801.2005.00130.x. PMID 16618333
- [Background] Lazar HL, McCann J, Fitzgerald CA, Cabral HJ. Adhesive strips versus subcuticular suture for mediansternotomy wound closure. J Card Surg. 2011 Jul;26(4):344-7. doi: 10.1111/j.1540-8191.2011.01257.x. Epub 2011 May 9. PMID 21554389
- [Background] Hall LT, Bailes JE. Using Dermabond for wound closure in lumbar and cervical neurosurgical procedures. Neurosurgery. 2005 Jan;56(1 Suppl):147-50; discussion 147-50. doi: 10.1227/01.neu.0000144170.39436.52. PMID 15799803
- [Background] Asomugha EU, Miller JA, McLain RF. Surgical Site Infections in Posterior Lumbar Surgery: A Controlled-Cohort Study of Epidural Steroid Paste. Spine (Phila Pa 1976). 2017 Jan 1;42(1):63-69. doi: 10.1097/BRS.0000000000001668. PMID 27135641
- [Background] Saeedinia S, Nouri M, Azarhomayoun A, Hanif H, Mortazavi A, Bahramian P, Yarandi KK, Amirjamshidi A. The incidence and risk factors for surgical site infection after clean spinal operations: A prospective cohort study and review of the literature. Surg Neurol Int. 2015 Sep 29;6:154. doi: 10.4103/2152-7806.166194. eCollection 2015. PMID 26500800